CLINICAL TRIAL: NCT06042335
Title: A Feasibility Study for the DAISe EZ Thrombectomy Device - Pacific
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MIVI Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102699
Record Dates: First submitted 2023-08-25; First posted 2023-09-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- DAISe EZ (Experimental): Mechanical thrombectomy utilizing the DAISe Thrombectomy System, consisting of the DAISe Thrombectomy Device and DAISe Delivery Catheter, used with aspiration.
  Interventions: Device: DAISe EZ

INTERVENTIONS:
Device: DAISe EZ — DAISe Thrombectomy System for mechanical thrombectomy

SUMMARY:
The study is a prospective, multi-center, single arm, feasibility study that will enroll a maximum of 20 subjects. A maximum of 5 investigational centers in Australia will participate. Enrollment is expected to take about 4 months, subject participation will last about 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Pre-stroke (24 hours prior to stroke onset) independent functional status in activities of daily living with modified Rankin Score 0-2.
3. Diagnosis of acute ischemic stroke with study enrollment time < 24 hours from onset of symptoms.
4. Disabling stroke defined as a baseline NIHSS > 6.
5. Confirmed symptomatic, large vessel occlusion of the intracranial internal carotid artery (ICA), MCA-M1 or MCA-M2.
6. The following imaging criteria must also be met:

   * For subjects 0-6hrs onset:

     * MRI criterion: volume of diffusion restriction as assessed by automated core volume software ≤50 mL OR
     * CT criterion: ASPECTS 6 to 10 on baseline CT or CTA-source images or, computed tomography perfusion (CPT) core as assessed by automated core volume software ≤50 mL.
   * For subjects 6-24hrs onset:

     * ≤20mL ischemic core volume if age >80
     * ≤30mL ischemic core volume if age <80 and NIHSS 10-20
     * ≤50mL ischemic core volume if age <80 and NIHSS >20
7. Signed informed consent from patient or legal representative

Exclusion Criteria:

1. Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage on presentation.
2. Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic.
3. Rapidly improving neurological deficits based on the investigator's clinical judgement.
4. Pregnancy; if a woman is of child-bearing potential and urine or serum beta HCG test is positive.
5. Severe contrast allergy or absolute contraindication to iodinated contrast.
6. Difficult endovascular access, difficult aortic arch or severe neurovascular tortuosity that will result in an inability to deliver endovascular therapy.
7. Evidence of dissection in the carotid or target artery for treatment.
8. Presence of a carotid artery stenosis or occlusion requiring balloon angioplasty or stenting at time of the procedure.
9. Renal failure (on dialysis).
10. Severe, sustained hypertension resistant to treatment (SBP >185 mmHg or DBP >110 mmHg).
11. Use of warfarin anticoagulation with International Normalized Ratio (INR) > 3.0 at the time of the procedure or any known hemorrhagic or coagulation deficiency.
12. Use of a direct thrombin inhibitor within the last 48 hours; partial thromboplastin time (PTT) > 2.0 times the normal prior to procedure.
13. Cerebral vasculitis or evidence of active systemic infection.
14. Suspicion of aortic dissection, presumed septic embolus or suspicion of bacterial endocarditis.
15. Clinical symptoms suggestive of bilateral stroke or occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
16. A severe or fatal comorbid illness that will prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Successful revascularization | Peri-Procedural
  Defined as proportion of subjects with mTICI 2b-3 flow post treatment with the DAISe Thrombectomy Device.
Symptomatic intracranial hemorrhage (sICH) at 24 hours post-procedure | 24 Hours [window: 12-36 hours] post procedure
  Defined as proportion of subjects with Symptomatic intracranial haemorrhage (sICH) at 24 hours post-procedure as detected by CT/MRI with clinical deterioration of an NIHSS change of greater than or equal to 4.

IPD SHARING:
Plan to Share IPD: No